CLINICAL TRIAL: NCT01526486
Title: Videoscopic Versus Open Inguinal Lymphadenectomy for Sentinel Node Positive Cutaneous Malignancies and Genitourinary Staging Procedures
Brief Title: Videoscopic Versus Open Inguinal Lymphadenectomy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Keith A Delman, MD, Associate Professor of Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012329; WCI1585-08 (Other: Winship Cancer Institute)
Record Dates: First submitted 2012-01-28; First posted 2012-02-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Melanoma; Merkel Cell Carcinoma; Squamous Cell Carcinoma; Penile Carcinoma; Urethral Carcinoma; Extramammary Paget's Disease; Scrotal Carcinoma; Anal Cancer; Vulvar Cancer; Skin Cancer; Lymphadenopathy
Keywords: melanoma; urology; inguinal; lymph nodes; groin; lymphadenectomy; groin dissection; skin cancer; penile cancer; urethral cancer; scrotal cancer; Paget's disease
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Carcinoma, Squamous Cell; Penile Neoplasms; Urethral Neoplasms; Paget Disease, Extramammary; Anus Neoplasms; Vulvar Neoplasms; Skin Neoplasms; Lymphadenopathy; Osteitis Deformans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videoscopic (Minimally invasive) (Experimental): Patients in this arm will have the procedure done through the three port minimally invasive approach.
  Interventions: Procedure: Videoscopic procedure
- Open (traditional approach) (Active Comparator): Patients in this arm will have the traditional, open approach in conjunction with a sartorius muscle transposition.
  Interventions: Procedure: Open, traditional approach

INTERVENTIONS:
Procedure: Videoscopic procedure — Minimally invasive, three port approach, (using a laparoscope to perform a procedure previously performed through open surgery).
  Arms: Videoscopic (Minimally invasive)
Procedure: Open, traditional approach — Open surgical procedure, with sartorius muscle transfer.
  Arms: Open (traditional approach)

SUMMARY:
Patients with melanoma, some other rare skin cancers, and some cancers of the penis and scrotum can have their cancer spread to the lymph nodes in the upper part of the leg, called the groin. Medically, this area is called the inguinal area. At present, for melanomas and skin cancers this type of spread is usually found with a special test called a "sentinel lymph node biopsy". This procedure can find spread of even a few cells in a single lymph node-allowing the treating doctor to find the spread very early.

Treatment for patients with skin cancer in the lymph nodes in this area is to remove all of the lymph nodes in this area. In patients with cancers of the penis and scrotum who do hot have any evidence of cancer having spread either by physical examination or by radiology tests, the lymph nodes in this area are removed to check and see if there is cancer in them. This is called staging.

At present, the standard way to remove all of the lymph nodes in the groin is by a large incision, approximately 8-10 inches in length. For patients who have this operation, there is a very high incidence of infection after surgery: as many as 50% as patients can have a problem after surgery. These infections range from a low grade skin infection needing oral antibiotics to deep infections requiring the wound to be opened and occasionally needing readmission to the hospital and antibiotics given via the vein.

With the advent of new technology and new equipment, the ability to perform this procedure through small incisions away from the groin and further down the leg has become possible. This procedure has never been performed routinely nor compared side by side to the standard open approach. The investigators propose to perform this protocol in two phases.

The investigators have performed procedures in 20 groins to this point and have confirmed the number of lymph nodes and visually verified that the procedure is identical to the open procedure. The investigators performed these procedures in order to insure that the investigators were offering an equivalent option regardless of which procedure the patient is randomized to.

The study will involve the randomization of patients undergoing the procedure. The investigators will randomize the next 110 patients in a 2:1 fashion (two people will get the videoscopic procedure for every one who gets the open procedure) until 73 patients are included in the video arm and 37 in the open arm. Outcomes including recurrence rate, duration of drain requirements, and incidence of lymphedema will be followed. Patients will be followed using standard of care processes, including regular office visits, physical exams, and radiographic imaging, when indicated. Patients will be followed for 5 years.

DETAILED DESCRIPTION:
Inguinal lymphadenectomy is the standard procedure used to treat patients with metastatic lymphadenopathy to the groin. For melanoma, the majority of these patients are diagnosed via sentinel lymph node biopsy, which identifies disease at a very early stage. In up to 80% of patients no additional disease is identified in the lymphadenectomy specimen1,2, which is performed at a separate setting from the initial biopsy, unlike in breast cancer. Unfortunately, due to the nature of the incision and the location, inguinal lymphadenectomy is associated with an extremely high incidence of postoperative wound complications. As many as 50% of patients will develop wound infections ranging from simple cellulitis to significant wound abscesses requiring a reopening of the incision and considerable wound care, sometimes necessitating rehospitalization.3 These data are associated with an open procedure, generally requiring a 10-15 cm incision. Recently, a videoscopic approach to this procedure has been described.4 It has been well-proven that a minimally invasive approach to cancer surgery does not have a negative impact on outcomes from cancer treatment.5 Emory has long been at the forefront of minimally invasive surgery and it is only appropriate that the investigators continue to lead the field. As one of the busiest melanoma centers in the country, the investigators have the opportunity to demonstrate the utility of this approach and continue to lead the field in both cancer therapy and minimally invasive surgery.

The trial will randomize patients to either videoscopic or open lymphadenectomy to determine if there is any difference in wound complication rate and as a secondary endpoint, time to recurrence. It is expected that there will be a substantial (approximately 25% incidence versus traditional 50% incidence or half of the number of wound complications) decrease in the incidence of wound complications after minimally invasive lymphadenectomy. This is expected predominantly for two reasons: 1. The wounds for this procedure are outside of the groin, in contrast being located on the thigh, a less difficult area for healing; and 2. The wounds are markedly shorter in length, making wound healing easier. The investigators would expect recurrence patterns to be identical in the two groups. The investigators have performed 20 procedures using the minimally invasive approach, and our experience to this point has demonstrated that the mean and median number of nodes harvested was 9 and 10.5 respectively. Median procedure duration has been 147 minutes and there have been 3 patients (15%) with complications (1 seroma, 2 with superficial cellulitis) but there have been no wound dehiscences or superficial breakdowns.

While the investigators do not have immediate access to the entire dataset of patients treated at Emory with the open approach, the investigators do have complete data on the 40 patients most recently treated (over the last 2 years). Of these 40 patients, 17 (43%) had complications other than lymphedema. Of these, 5 required hospitalization and two had complete wound dehiscences requiring management with a wound vacuum-assisted closure (VAC). This data is not complete, but reasonably reflects the Emory experience and allows us to conclude that our data is similar to that reported in the literature historically.

While many minimally invasive approaches to open procedures have been applied without randomized trials proving their efficacy (splenectomy, hepatectomy, pancreatectomy, partial gastrectomy, to name a few), the investigators believe it is prudent when adopting a new approach for a cancer operation to study it in a prospective fashion. This is the only trial of its kind and the investigators are one of only a few centers in the world that has the minimally invasive knowledge and expertise and the volume of urologic and melanoma patients to have the potential to perform such a trial. It is incumbent upon us to complete this study.

The goal of this study is to determine if a videoscopic approach to a standard procedure offers a better outcome for patients with respect to wound complications and to prove that there is no inferiority between the videoscopic approach and the traditional open approach from a cancer outcome standpoint, specifically time to recurrence and nodal yield.

Patients will be considered for this study if they are between age 18 and 80, have either metastatic melanoma or merkel cell carcinoma diagnosed by sentinel lymph node biopsy or have indications for inguinal lymphadenectomy for urological malignancy.

The study will be designed as a randomized, prospective trial, analyzing wound complications as the primary endpoint and recurrence-free survival as a secondary endpoint. Our sample size calculation (see section 8.0 below) indicate that a sample size of 73 patients in the study arm and 37 patients in the control arm will be sufficient to detect a moderate-to-strong effect with an 80% power and a 95% level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered for this study if they are between age 18 and 80
* Patients have either metastatic melanoma or merkel cell carcinoma diagnosed by sentinel lymph node biopsy or are candidates for a staging procedure for either a penile or scrotal carcinoma

Exclusion Criteria:

* Patients with unresectable metastatic disease
* Patients who are pregnant or lactating
* Patients with prohibitive cardiac or pulmonary comorbidities
* Patients with other contraindications for general anesthesia as determined by the anesthesia preoperative evaluation will not be considered enrolled in the trial although they may undergo randomization prior to exclusion from surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Complication profile | 30 days
  The primary objective is to assess wound infection, wound dehiscence and other wound complications.
Length of stay | 1- 7 days
  Hospital length of stay.
Lymphedema | 5 years
  Assessment of lymphedema will be determined in all patients to identify if there is a difference in all patients undergoing either videoscopic or open inguinal lymphadenectomy.
Nodal yield | 5-7 days post procedure
  This will characterize, as a surrogate of completeness of surgery, the number of nodes retrieved at the surgical procedure via either approach.

SECONDARY OUTCOMES:
Readmission | 30 days
  To assess differences in readmission rates between the two groups.
Oncologic outcomes--survival | 5 years
  Recurrence free and overall survival will be measured in patients undergoing the procedure to determine if the procedure impacts survival at all.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Delman, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital-Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Background] Delman KA, Kooby DA, Rizzo M, Ogan K, Master V. Initial experience with videoscopic inguinal lymphadenectomy. Ann Surg Oncol. 2011 Apr;18(4):977-82. doi: 10.1245/s10434-010-1490-5. Epub 2010 Dec 24. PMID 21184190
- [Background] Delman KA, Kooby DA, Ogan K, Hsiao W, Master V. Feasibility of a novel approach to inguinal lymphadenectomy: minimally invasive groin dissection for melanoma. Ann Surg Oncol. 2010 Mar;17(3):731-7. doi: 10.1245/s10434-009-0816-7. PMID 20183910
- [Background] Master V, Ogan K, Kooby D, Hsiao W, Delman K. Leg endoscopic groin lymphadenectomy (LEG procedure): step-by-step approach to a straightforward technique. Eur Urol. 2009 Nov;56(5):821-8. doi: 10.1016/j.eururo.2009.07.003. Epub 2009 Jul 15. PMID 19640633
- [Background] Tobias-Machado M, Tavares A, Molina WR Jr, Zambon JP, Medina JA, Forseto PH Jr, Juliano RV, Wroclawski ER. Video endoscopic inguinal lymphadenectomy (VEIL): initial case report and comparison with open radical procedure. Arch Esp Urol. 2006 Oct;59(8):849-52. doi: 10.4321/s0004-06142006000800020. PMID 17153511
- See also: Link to Dr. Delman's Profile page — https://winshipcancer.emory.edu/bios/faculty/delman-keith.html
- See also: Link to Dr. Master's Profile Page — https://winshipcancer.emory.edu/bios/faculty/master-viraj.html